CLINICAL TRIAL: NCT01302691
Title: A Phase III, Randomized, Active-Comparator Controlled Clinical Trial to Study the Efficacy and Safety of MK-0954E in Japanese Patients With Essential Hypertension Uncontrolled With Losartan and Amlodipine Co-administration
Brief Title: MK-0954E Study in Participants With Hypertension (MK-0954E-357)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0954E-357
Record Dates: First submitted 2011-02-22; First posted 2011-02-24 (Estimated); Results first posted 2017-01-27 (Estimated); Last update posted 2019-03-15 (Actual); Status verified 2019-02

CONDITIONS: Hypertension
Keywords: Essential hypertension; Uncontrolled hypertension; Antihypertensive agents; Blood pressure
MeSH Terms: conditions — Hypertension; Essential Hypertension | interventions — Losartan; Hydrochlorothiazide; Amlodipine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- L50/H12.5/A5 (Experimental): Participants receive 1 tablet, containing 50 mg losartan potassium (L50), 12.5 mg hydrochlorothiazide (H12.5), and 5 mg amlodipine besylate (A5), orally, once daily, for 8 weeks.
  Interventions: Drug: losartan potassium + hydrochlorothiazide + amlodipine besylate (MK-0954E); Drug: Placebo to losartan potassium; Drug: Placebo to amlodipine besylate
- L50 + A5 (Active Comparator): Participants receive tablet, containing 50 mg losartan potassium (L50), and tablet containing 5 mg amlodipine besylate (A5), orally, once daily, for 8 weeks.
  Interventions: Drug: Losartan potassium; Drug: Amlodipine besylate; Drug: Placebo to MK-0954E

INTERVENTIONS:
Drug: losartan potassium + hydrochlorothiazide + amlodipine besylate (MK-0954E) — One tablet, containing 50 mg losartan potassium, 12.5 mg hydrochlorothiazide, and 5 mg amlodipine besylate, orally, once daily, for 8 weeks.
  Arms: L50/H12.5/A5
Drug: Losartan potassium — One tablet, containing 50 mg losartan potassium, orally, once daily, for 8 weeks.
  Arms: L50 + A5
Drug: Amlodipine besylate — One capsule, containing 5 mg amlodipine besylate, orally, once daily, for 8 weeks.
  Arms: L50 + A5
Drug: Placebo to MK-0954E — One tablet, containing placebo, orally, once daily, for 8 weeks.
  Arms: L50 + A5
Drug: Placebo to losartan potassium — One tablet, containing placebo, orally, once daily, for 8 weeks.
  Arms: L50/H12.5/A5
Drug: Placebo to amlodipine besylate — One capsule, containing placebo, orally, once daily, for 8 weeks.
  Arms: L50/H12.5/A5

SUMMARY:
This study is being done to evaluate the efficacy, safety, and tolerability of losartan potassium 50 mg (L50) + hydrochlorothiazide 12.5 mg (H12.5) + amlodipine besylate 5 mg (A5) (MK-0954E). The primary hypothesis is that L50/H12.5/A5 is more effective in lowering mean trough sitting diastolic blood pressure (SiDBP) after 8 weeks of treatment compared to L50+A5 in Japanese participants with essential hypertension who are not adequately controlled following an 8-week treatment with filter period study drug (L50+A5).

ELIGIBILITY:
Inclusion criteria

* Participant has a diagnosis of essential hypertension.
* Participant is being treated with single or dual treatment for hypertension and will be able to discontinue the prior antihypertensive medication.
* Participant has a mean trough SiDBP of ≥ 90 mmHg and < 110 mmHg.
* Participant has a mean trough SiSBP of ≥ 140 mmHg and < 200 mmHg.
* Participant has no clinically significant abnormality at screening visit.

Exclusion criteria

* Participant is currently taking > 2 antihypertensive medications.
* Participant has a history of significant multiple and/or severe allergies to ingredients of Nu-Lotan or Preminent, amlodipine or dihydropyridine drug, and thiazide drug or related drug (i.e., sulfonamide-containing "chlortalidone" medicines).
* Participant is, at the time of signing informed consent, a user of recreational or illicit drugs or has had a recent history within the last year of drug or alcohol abuse or dependence.
* Participant is pregnant or breastfeeding, or expecting to conceive OR the pregnancy test is positive at screening visit (Visit 1).
* Participant is currently participating or has participated in a study with an investigational compound or device within 30 days of signing informed consent.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 327 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2012-04-01 (Actual); Study Completion 2012-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Rakugi H, Tsuchihashi T, Shimada K, Numaguchi H, Nishida C, Yamaguchi H, Shirakawa M, Azuma K, Fujita KP. Efficacy and safety of fixed-dose losartan/hydrochlorothiazide/amlodipine combination versus losartan/hydrochlorothiazide combination in Japanese patients with essential hypertension. Clin Exp Hypertens. 2015;37(3):260-6. doi: 10.3109/10641963.2014.954712. Epub 2014 Oct 1. PMID 25271811
- [Result] Rakugi H, Tsuchihashi T, Shimada K, Numaguchi H, Nishida C, Yamaguchi H, Shirakawa M, Azuma K, Fujita KP. Add-on effect of hydrochlorothiazide 12.5 mg in Japanese subjects with essential hypertension uncontrolled with losartan 50 mg and amlodipine 5 mg. Hypertens Res. 2015 May;38(5):329-35. doi: 10.1038/hr.2015.3. Epub 2015 Feb 26. PMID 25716649

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All participants received single-blind losartan 50 mg (L50) + amlodipine 5 mg (A5) and placebo for L50/(H12.5)/A5 during 8-week Filter/Screening Period. A total of 707 entered the Filter/Screening Period and 327 were randomly assigned to 1 of the 2 treatment arms for the Double-blind Treatment Period.
Period: Overall Study
Arm/Group | L50/H12.5/A5 | L50 + A5
Started | 164 | 163
Completed | 154 | 157
Not Completed | 10 | 6
Not completed — Adverse Event | 2 | 0
Not completed — Death | 0 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Blood Pressure/Potassium Criteria Met | 6 | 4
Not completed — Physician Decision | 0 | 1
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | L50/H12.5/A5 | L50 + A5 | Total
Number analyzed (Participants) | 164 | 163 | 327
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.9 (9.4) | 55.4 (10.1) | 55.2 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 41 | 74
  Male | 131 | 122 | 253

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Trough Sitting Diastolic Blood Pressure (SiDBP)
Description: Sitting diastolic blood pressure was measured by automated sphygmomanometer pre-dose on Day 1 (baseline) and at 24 ± 2 hours after the last study drug administration at Week 8. The difference between the baseline and Week 8 assessments was calculated and summarized by treatment arm.
Time Frame: Baseline and Week 8
Population: All participants that received at least one dose of study treatment, had at least 1 post-randomization observation for the analysis endpoint, and had baseline data
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Arm/Group | L50/H12.5/A5 | L50 + A5
Number analyzed (Participants) | 164 | 163
mmHg | -9.1 [-10.2 to -7.9] | -8.0 [-9.1 to -6.8]
Statistical Analysis 1: Comparison: L50/H12.5/A5 vs L50 + A5; Test type: Superiority or Other; p = 0.205, Constrained Longitudinal Data Analysis; Model includes treatment group, time point, and the interaction of time by treatment with restriction of same baseline mean across treatment groups; Difference in Least Squares Means = -1.1, 95% CI 2-sided [-2.7 to 0.6]

2. Primary Outcome: Percentage of Participants Who Experience ≥1 Adverse Event (AE)
Description: An AE was defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the product, whether or not considered related to the use of the product. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition which was temporally associated with the use of the product, was also an AE. The percentage of participants who experienced at least 1 AE during the 10-week treatment and follow-up period were summarized by study drug received.
Time Frame: up to 14 days after last dose of study drug (up to 10 weeks)
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: Percentage of Participants
Arm/Group | L50/H12.5/A5 | L50 + A5
Number analyzed (Participants) | 164 | 163
Percentage of Participants | 30.5 | 28.8

3. Primary Outcome: Percentage of Participants Who Experience ≥1 Drug-related AE
Description: An AE was defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the product, whether or not considered related to the use of the product. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition which was temporally associated with the use of the product, was also an AE. Percentage of participants that experienced at least 1 AE that was reported as possibly, probably, or definitely related to the study drug by the investigator during the 10-week treatment and follow-up period were summarized by study drug received.
Time Frame: up to 14 days after last dose of study drug (up to 10 weeks)
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: Percentage of Participants
Arm/Group | L50/H12.5/A5 | L50 + A5
Number analyzed (Participants) | 164 | 163
Percentage of Participants | 11.6 | 3.7

4. Primary Outcome: Percentage of Participants Who Experience ≥1 Serious Adverse Event (SAE)
Description: An SAE is any AE occurring at any dose or during any use of Sponsor's product that does the following: results in death; is life threatening; results in persistent or significant disability/incapacity; results in or prolongs an existing inpatient hospitalization; is a congenital anomaly/birth defect; is a cancer; is associated with an overdose; is another important medical event. The percentage of participants who experienced at least 1 SAE during the 10-week treatment and follow-up period were summarized by study drug received.
Time Frame: up to 14 days after last dose of study drug (up to 10 weeks)
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: Percentage of Participants
Arm/Group | L50/H12.5/A5 | L50 + A5
Number analyzed (Participants) | 164 | 163
Percentage of Participants | 0.6 | 0.6

5. Primary Outcome: Percentage of Participants Who Experience ≥1 Drug-related SAE
Description: An SAE is any AE occurring at any dose or during any use of Sponsor's product that does the following: results in death; is life threatening; results in persistent or significant disability/incapacity; results in or prolongs an existing inpatient hospitalization; is a congenital anomaly/birth defect; is a cancer; is associated with an overdose; is another important medical event. Percentage of participants that experienced at least 1 SAE that was reported as possibly, probably, or definitely related to the study drug by the investigator during the 10-week treatment and follow-up period were summarized by study drug received
Time Frame: up to 14 days after last dose of study drug (up to 10 weeks)
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: Percentage of Participants
Arm/Group | L50/H12.5/A5 | L50 + A5
Number analyzed (Participants) | 164 | 163
Percentage of Participants | 0.0 | 0.0

6. Primary Outcome: Percentage of Participants Who Had Study Drug Stopped Due to an AE
Description: An AE was defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the product, whether or not considered related to the use of the product. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition which was temporally associated with the use of the product, was also an AE. The percentage of participants who had study drug stopped during the 8-week treatment period due to an AE regardless of whether or not they completed the study was summarized by treatment arm
Time Frame: up to 8 weeks
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: Percentage of Participants
Arm/Group | L50/H12.5/A5 | L50 + A5
Number analyzed (Participants) | 164 | 163
Percentage of Participants | 1.2 | 0.0

7. Secondary Outcome: Change in Mean Trough Sitting Systolic Blood Pressure (SiSBP)
Description: Sitting systolic blood pressure was measured by automated sphygmomanometer pre-dose on Day 1 (baseline) and at 24 ± 2 hours after the last study drug administration at Week 8. The difference between the baseline and Week 8 assessments was calculated and summarized by treatment arm.
Time Frame: Baseline and Week 8
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Arm/Group | L50/H12.5/A5 | L50 + A5
Number analyzed (Participants) | 164 | 163
mmHg | -13.4 [-15.2 to -11.6] | -10.2 [-12.0 to -8.4]
Statistical Analysis 1: Comparison: L50/H12.5/A5 vs L50 + A5; Test type: Superiority or Other; p = 0.011, Constrained Longitudinal Data Analysis; [statistical method as in outcome 1, analysis 1]; Difference in Least Squares Means = -3.2, 95% CI 2-sided [-5.7 to -0.8]

ADVERSE EVENTS:
Time Frame: up to 2 weeks after last dose of study drug (up to 10 weeks)
Description: All participants that received at least 1 dose of study drug.
Arm/Group | L50/H12.5/A5 | L50 + A5
Serious Adverse Events (participants affected / at risk) | 1/164 | 1/163
Other Adverse Events (participants affected / at risk) | 11/164 | 15/163
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | L50/H12.5/A5 (N=164) | L50 + A5 (N=163)
Sudden cardiac death (General disorders) | 0 (0) | 1 (1)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | L50/H12.5/A5 (N=164) | L50 + A5 (N=163)
Nasopharyngitis (Infections and infestations) | 11 (11) | 15 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission. Sponsor review can be expedited to meet publication timelines.